CLINICAL TRIAL: NCT06632600
Title: A Randomized, Participant- and Investigator-blinded, Controlled, Parallel Group Study to Assess the Efficacy, Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LXE408 in Participants With Chronic Chagas Disease Without Severe Organ Dysfunction.
Brief Title: A Study of Efficacy, Safety, Tolerability of LXE408 in Participants With Chronic Chagas Disease.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLXE408B12201
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Chagas Disease
Keywords: LXE408; Chronic Chagas disease; Chronic indeterminate Chagas disease; Chronic Chagas disease without severe organ dysfunction; CICD; Chronic CD; Trypanosoma cruzi
MeSH Terms: conditions — Chagas Disease | interventions — LXE408; benzonidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The benznidazole arm is open-label.
  For the LXE and placebo arms:
  Participants, investigator, staff, and persons performing the assessments will remain blinded to the identity of the treatment from the time of randomization until 12 month database lock for blinded arms. The sponsor clinical trial team (CTT) will be blinded until the primary endpoint analysis (when all participants complete 6 month visit) and may become unblinded as needed at any other interim analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LXE408 28 days (Experimental): LXE408 administered by oral route
  Interventions: Drug: LXE408
- LXE408 14 days and Placebo 14 days (Experimental): LXE408 administered by oral route, followed by Placebo administered by oral route
  Interventions: Drug: LXE408; Drug: Placebo
- Placebo 28 days (Placebo Comparator): Placebo administered by oral route
  Interventions: Drug: Placebo
- Benznidazole 60 days (Active Comparator): Benznidazole administered by oral route
  Interventions: Drug: Benznidazole

INTERVENTIONS:
Drug: LXE408 — LXE408 administered by oral route
  Arms: LXE408 14 days and Placebo 14 days; LXE408 28 days
Drug: Placebo — Placebo administered by oral route
  Arms: LXE408 14 days and Placebo 14 days; Placebo 28 days
Drug: Benznidazole — Benznidazole administered by oral route (administered as standard of care)
  Arms: Benznidazole 60 days

SUMMARY:
This study is to investigate the ability of LXE408 to clear or reduce the level of parasites in the blood of people with chronic Chagas disease. Participants must have chronic Chagas disease without severe organ dysfunction.

DETAILED DESCRIPTION:
This is an interventional, phase 2, PoC (Proof of Concept) randomized, participant- and investigator-blinded, controlled, parallel group study, with 4 treatment arms. The purpose of this study is to assess the efficacy (anti-parasitological activity), safety, PK (pharmacokinetics), and PD (pharmacodynamics) of LXE408 in participants with CICD (chronic indeterminate Chagas disease) and chronic Chagas disease without severe cardiac or gastrointestinal dysfunction compared to placebo and to benznidazole.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged ≥ 18 years to ≤ 60 years old
* Confirmed diagnosis of T. cruzi infection
* History that participant has been determined to be in chronic phase of CD
* Written informed consent must be obtained before any assessment is performed, and participants should express understanding of the consent form and the study
* Participants must be considered by the investigator eligible for and able to comply with local prescribing information for benznidazole
* Ability and willingness to communicate well with the investigator/study site and comply with requirements of the study

Exclusion Criteria:

* Signs (on physical examination) and/or symptoms of CD in the acute phase as determined by the investigator at screening
* History of CD treatment with benznidazole or nifurtimox at any time in the past
* History of and/or current (at screening) symptoms or signs (physical examination findings) of moderate or severe CD-related gastrointestinal disease
* Participants who weigh < 50 kg or >90kg at screening
* At sites conducting the MRI assessments, participants may participate in the overall study, but will be excluded from the MRI assessment if they have contraindications to MRI imaging
* Any clinically significant disease during screening that, in the opinion of the investigator, would put the safety of the participant at risk through participating, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study, or would compromise participant compliance or preclude completion of the study
* Documented history or current findings at screening of clinically significant cardiovascular conditions such as, but not limited to: unstable ischemic heart disease; NYHA Class III/IV heart failure (due to Chagas disease or other conditions); arrhythmias
* Known or suspected ongoing, chronic or recurrent viral, bacterial or fungal infectious diseases including but not limited to: Tuberculosis, leishmaniasis, severe malaria, atypical mycobacterial infection, listeriosis, aspergillosis, or endemic mycoses, and/or documented positivity for human immunodeficiency virus (HIV) infection.

  * Participants with controlled HIV on antiretroviral therapy are eligible to participate if CD4 ≥ 500 at screening
* History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system within the past 5 years prior to screening (except for basal cell carcinoma or actinic keratosis that have been treated with no evidence of recurrence in the past 3 months, carcinoma in situ of the cervix or non-invasive malignant colon polyps that have been removed)
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the participant during the study period

  * Pancreatic injury or pancreatitis: If any single parameter of amylase or lipase exceeds 1.5x ULN at screening Participants with known recurrent pancreatitis (more than 1 episode in lifetime, from any cause) are excluded
  * Liver disease or liver injury as indicated by abnormal liver function tests (LFTs):

Any single parameter of ALT, AST, alkaline phosphatase must not exceed 1.5x ULN at screening Serum bilirubin must not exceed the ULN at screening elevated serum bilirubin is not excluded if there is a documented history of Gilbert's Syndrome

* History of renal disease as indicated by creatinine level above 1.5x ULN or microalbuminuria at screening; Evidence of urinary obstruction, or difficulty in voiding at screening; evidence of congenital renal abnormalities with known effect on renal function; calculated eGFR <60 mL/min (<0.835 mL/s) using the CKD-EPI formula for adults

  * Participants with screening hematology parameters outside of the thresholds
  * Current use of medications prohibited by the protocol at screening and/or baseline visits, or expected use of any prohibited medication during the study treatment period
* Use of benznidazole in the blinded arms is prohibited until unblinding occurs after all participants complete Month 12.

  * Use of other investigational drugs at the time of study drug dosing
  * History of multiple and recurring allergies or allergy to the investigational compound/compound class being used in this study or to benznidazole
  * History of drug abuse or unhealthy alcohol use within the 12 months prior to dosing
  * Pregnant or nursing (lactating/breast-feeding) women
  * Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 5 days after stopping of investigational drug and benznidazole
  * Participants who, in the opinion of the investigator, will not be able to comply with study procedures or visits, adhere to dosing schedule, or other otherwise be in compliance with study requirements

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2027-03-22 (Estimated); Study Completion 2030-09-21 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of sustained parasitological clearance using polymerase chain reaction (PCR) results over 6 months - LXE408 28 days versus placebo. | At Months 2, 4, and 6
  The parasitological load will be measured using polymerase chain reaction (PCR) at 2 months, 4 months, and at 6 months. At each timepoint, multiple samples are evaluated. The participant will be considered negative at a visit if the parasite is not detectable in all samples at a visit and positive if the parasite level is detectable in at least one sample. Sustained parasitological clearance is achieved if participant is negative at all 3 visits.

SECONDARY OUTCOMES:
Presence or absence of sustained parasitological clearance using polymerase chain reaction (PCR) results over 6 months - LXE408 -14 days versus placebo | At Months 2, 4, and 6
  The parasitological load will be measured using polymerase chain reaction (PCR) at 2 months, 4 months, and at 6 months. At each timepoint, multiple samples are evaluated. The participant will be considered negative at a visit if the parasite is not detectable in all samples at a visit and positive if the parasite level is detectable in at least one sample. Sustained parasitological clearance is achieved if participant is negative at all 3 visits.
Presence or absence of sustained parasitological clearance using polymerase chain reaction (PCR) results over 6 months-LXE408 - 28 days and 14 days versus benznidazone | At Months 2, 4, and 6
  The parasitological load will be measured using polymerase chain reaction (PCR) at 2 months, 4 months, and at 6 months. At each timepoint, multiple samples are evaluated. The participant will be considered negative at a visit if the parasite is not detectable in all samples at a visit and positive if the parasite level is detectable in at least one sample. Sustained parasitological clearance is achieved if participant is negative at all 3 visits.
Presence or absence of early parasitological clearance | At Day 7, 14 and 28
  The parasitological load will be measured using polymerase chain reaction (PCR). The participant will be considered negative at a visit if the parasite is not detectable in all samples at a visit and positive if the parasite level is detectable in at least one sample.
Presence or absence of sustained parasitological clearance over 12 months by PCR testing | 12 Months
  The parasitological load will be measured using polymerase chain reaction (PCR). The participant will be considered negative at a visit if the parasite is not detectable in all samples at a visit and positive if the parasite level is detectable in at least one sample. Sustained parasitological clearance is achieved if participant is negative at all subsequent visits.
Time to parasitological clearance based on serial PCR testing | 12 Months
  Time to parasitological clearance based on PCR by treatment will be estimated using the Kaplan-Meier approach.
Presence or absence of seroreversion using conventional serology | At Month 6 and Month 12
  Seroreversion as measured by conventional serology will be evaluated at 6 and 12-month study visits. Seroreversion is determined by the proportion of participants achieving serology changes from positive at baseline to negative at each time point.
Occurrence and severity of treatment emergent adverse events during the study | Up to 12 Months
  Incidence and severity of AEs by treatment group, including changes in the vital signs, electrocardiogram and laboratory results qualifying and reported as AEs.
Occurrence of adverse events resulting in treatment discontinuation | Up to 12 Months
  Incidence of AEs that result in treatment discontinuation.
Occurrence of all-cause mortality through end of study visit | Up to 48 Months
  Incidence of death through the end of study visit.
Maximum plasma concentration (Cmax) of LXE408 | At Day 1, 7, 14, 28
  Cmax is defined as the maximum (peak) observed concentration following a dose.
Time to maximum plasma concentration (Tmax) of LXE408 | At Day 1, 7, 14, 28
  Tmax is defined as the time to reach maximum (peak) concentration following a dose.
Area under the plasma concentration-time curve from time 0 to 8 hours post-dose (AUC0-8) | At Day 1, 7, 14, 28
  AUC0-8 will be calculated by non-compartmental methods based on LXE408 plasma concentration data.
Pre-dose concentration | At Day 14 and Day 28
  Pre-dose concentration is the observed plasma concentration that is just prior to the beginning of, or at the end of a dosing interval.

CONTACTS AND LOCATIONS:
Locations (16):
- United States (4):
  - Olive View UCLA Educ and Res Ins, Sylmar, California
  - University of Florida Shands, Gainesville, Florida
  - Boston Medical Center, Boston, Massachusetts
  - Baylor College of Medicine, Houston, Texas
- Argentina (4):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Corrientes
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Formosa
- Brazil (3):
  - Novartis Investigative Site, Montes Claros, Minas Gerais
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, São Caetano do Sul, São Paulo
- Colombia (5):
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Yopal, Casanare Department
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Floridablanca
  - Novartis Investigative Site, San Gil

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Novartis.aspx